CLINICAL TRIAL: NCT03434600
Title: Comparison of the Oxford Unicompartmental Knee Prosthesis With the Sigma High Performance Partial Knee Using Rontgen Stereophotogrammetric Analysis in Patients With Primary Medial Unicompartmental Knee Osteoarthritis.
Brief Title: Comparison of Oxford UKA and Sigma UKA With RSA.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Regional Hospital Holstebro (Other)
Responsible Party: Principal Investigator, Daan Koppens, MD, Regional Hospital Holstebro
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HolstebroH
Record Dates: First submitted 2018-02-09; First posted 2018-02-15 (Actual); Last update posted 2019-05-20 (Actual); Status verified 2019-05

CONDITIONS: Knee Osteoarthritis; Knee Replacement; RSA
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Oxford (Active Comparator): Patients receiving an Oxford UKA, which is the standard treatment for patients with medial osteoarthritis of the knee at our department.
  Interventions: Other: Oxford UKA vs Sigma UKA
- Sigma (Experimental): Patients receiving a Sigma UKA, which is the experimental treatment.
  Interventions: Other: Oxford UKA vs Sigma UKA

INTERVENTIONS:
Other: Oxford UKA vs Sigma UKA

SUMMARY:
Comparison of two unicompartmental knee arthroplasties (UKA), to see if Sigma UKA performs equally good as the Oxford UKA. The study focuses on how well the arthroplasty is fixated to the bone and on the difference in wear of the plastic insert. Finally, the functional outcome after surgery is compared between the two arthroplasties.

Hypothesis:

H1: The Sigma UKA has an equal migration pattern compared to the Oxford UKA with a follow up of two years - that is, no significant difference in migration between 1-2 years follow-up.

H2: The Oxford and Sigma UKA's have comparable polyethylene wear with a follow up of 5 years.

H3: The Oxford and Sigma UKA's have comparable patient perceived outcome measures (PROM) and leg extension power (LEP) postoperative.

H4: BMD of the proximal tibia does not influence migration of the tibial component

ELIGIBILITY:
Inclusion Criteria:

* All eligable patients with medial osteoarthritis of the knee.

Exclusion Criteria:

* - Inflammatory arthritis.
* Patients who are not able to participate in the fast-track surgery program.
* Patients with a contralateral knee arthroplasty.
* Patients who are unable to provide informed consent.
* Disseminated malignant disease (cancer) and treatment with radiation or chemotherapy.
* Serious systemic disease (e.g.. hemiparesis and severe parkinsonism)
* On-going case involving work injury of the knee.
* Female patients with a wish of becoming pregnant in the study period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Migration of prosthesis | 2 years follow-up
  RSA

SECONDARY OUTCOMES:
Bone mineral density | 2 years follow-up
  DXA
Polyethylene wear | 5 years follow-up
  Weight-bearing RSA

CONTACTS AND LOCATIONS:
Overall Officials: Daan Koppens, Principal Investigator — Hospital Unit Vest

IPD SHARING:
Plan to Share IPD: No